CLINICAL TRIAL: NCT00727857
Title: A Phase 3b, Double-Blind, Randomized Study to Determine the Efficacy and Safety of Pioglitazone HCl and Metformin HCl Fixed-Dose Combination Therapy Compared to Pioglitazone HCl Monotherapy and to Metformin HCl Monotherapy in the Treatment of Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety of Pioglitazone and Metformin Combination Therapy in Treating Type 2 Diabetes Mellitus.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-06-TL-OPIMET-008; U1111-1114-0371 (Registry Identifier: WHO)
Record Dates: First submitted 2008-07-30; First posted 2008-08-04 (Estimated); Results first posted 2010-03-09 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pioglitazone 15 mg /Metformin 850 mg BID (Experimental)
  Interventions: Drug: Pioglitazone and metformin
- Pioglitazone 15 mg BID (Active Comparator)
  Interventions: Drug: Pioglitazone
- Metformin 850 mg BID (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Pioglitazone and metformin — Pioglitazone 15 mg /metformin 850 mg combination, tablets, orally, twice daily for up to 24 weeks.
  Other Names: ACTOPLUS MET
  Arms: Pioglitazone 15 mg /Metformin 850 mg BID
Drug: Pioglitazone — Pioglitazone 15 mg, tablets, orally, twice daily for up to 24 weeks.
  Other Names: ACTOS®; AD4833
  Arms: Pioglitazone 15 mg BID
Drug: Metformin — Metformin 850 mg, tablets, orally, twice daily for up to 24 weeks.
  Other Names: Fortamet; Glucophage; Glucophage XR; Glumetza; Riomet
  Arms: Metformin 850 mg BID

SUMMARY:
The purpose of this study is to determine the efficacy of pioglitazone, twice daily (BID), combined with metformin versus pioglitazone taken alone and metformin taken alone in treating Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
Pioglitazone hydrochloride (ACTOS®) is a member of a class of oral antidiabetic agents known as thiazolidinediones, which act by reducing insulin resistance. Insulin resistance is a key feature of dysmetabolic syndrome and has been suggested to be the common pathophysiologic basis of both atherosclerosis and type 2 diabetes. Pioglitazone binds to peroxisome proliferator-activated receptors, an effect that is associated with altered transcription of genes capable of influencing carbohydrate and lipid metabolism.

Metformin hydrochloride is an oral antihyperglycemic drug not chemically or pharmacologically related to thiazolidinediones. Metformin is a biguanide, which has been shown to be effective in improving glycemic control in diabetic patients. Metformin inhibits hepatic glucose production, most likely through an inhibition of gluconeogenesis, and its use is associated with an improvement in tissue sensitivity to insulin. In accordance with published algorithms for the use of combination therapy for the treatment of type 2 diabetes, physicians have traditionally combined metformin with other antidiabetic agents.

This study will determine the effect of a fixed-dose combination of metformin with pioglitazone, compared to metformin monotherapy and pioglitazone monotherapy.

Study participation is anticipated to be approximately 6.5 months.

ELIGIBILITY:
Inclusion Criteria

* Has type 2 diabetes.
* Has received no treatment with antidiabetic medication in the 12 weeks prior to Screening, other than short-term use defined as less than or equal to 15 days.
* A glycosylated hemoglobin greater than or equal to 7.5% and less than or equal to 10.0% at Screening.
* Body mass index less than or equal to 45 kg/m2.
* Has received counseling on lifestyle modification for type 2 diabetes, including diet and exercise.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Stable condition as determined by a physician.

Exclusion Criteria

* Type 1 diabetes.
* Unstable angina or heart failure of any etiology with New York Heart Association functional class III or IV.
* History of myocardial infarction, cerebrovascular accident, percutaneous coronary intervention, coronary artery bypass graft, or transient ischemic attack in the 6 months prior to Screening.
* Male participant has a serum creatinine level greater than or equal to 1.5 mg per dL or female subject has a serum creatinine level greater than or equal to 1.4 mg per dL.
* Has a triglyceride level greater than 500 mg per dL.
* Male participant has a hemoglobin level less than 10.5 g per dL or female subject has a hemoglobin level less than 10.0 g per dL.
* Alanine aminotransferase level of greater than 2.5 times the upper limit of normal, active liver disease, or jaundice.
* History of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 2 alcoholic drinks per day) within 2 years prior to Screening.
* Has been discontinued from a thiazolidinedione or metformin therapy due to lack of efficacy or clinical or laboratory signs of intolerance.
* Previous history of cancer, other than basal cell or stage 1 squamous cell carcinoma, that has not been in remission for at least 5 years prior to the first dose of study medication.
* History of acute or chronic metabolic acidosis, including diabetic ketoacidosis with or without coma.
* Any disease or condition at Screening or Randomization that would compromise safety, might affect life expectancy, or make it difficult to successfully manage and follow the subject according to the protocol.
* Currently participating in another investigational study or has participated in an investigational study within 30 days prior to randomization.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Antidiabetic medications other than study medication
  * Chronically used oral or parenteral glucocorticoids
  * Niacin greater than 200 mg per day, including niacin-containing products such as Advicor
  * Chronically used steroid-joint injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science Strategy, Study Director — Takeda
Locations (77):
- United States (66):
  - Birmingham, Alabama
  - Haleyville, Alabama
  - Montgomery, Alabama
  - Pell City, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Artesia, California
  - Dinuba, California
  - Long Beach, California
  - Los Angeles, California
  - Norwalk, California
  - Orange, California
  - Santa Ana, California
  - Santa Monica, California
  - Pueblo, Colorado
  - Altamonte Springs, Florida
  - Coral Gables, Florida
  - Hialeah, Florida
  - Miami, Florida
  - Panama City, Florida
  - Plantation, Florida
  - Saint Cloud, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Columbus, Georgia
  - Boise, Idaho
  - Coeur d'Alene, Idaho
  - Chicago, Illinois
  - Flossmoor, Illinois
  - Peoria, Illinois
  - Elkhart, Indiana
  - Shawnee, Kansas
  - Southfield, Michigan
  - Chesterfield, Missouri
  - Billings, Montana
  - Elizabeth, New Jersey
  - Fayetteville, New York
  - New York, New York
  - Durham, North Carolina
  - Pinehurst, North Carolina
  - Cincinnati, Ohio
  - Perrysburg, Ohio
  - Zanesville, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Fleetwood, Pennsylvania
  - Norristown, Pennsylvania
  - Cranston, Rhode Island
  - Simpsonville, South Carolina
  - Varnville, South Carolina
  - Fayetteville, Tennessee
  - Corpus Christi, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Houston, Texas
  - McAllen, Texas
  - Mission, Texas
  - New Braunfels, Texas
  - North Richland Hills, Texas
  - San Antonio, Texas
  - Bountiful, Utah
  - Salt Lake City, Utah
  - Petersburg, Virginia
  - Port Orchard, Washington
  - Spokane, Washington
- Chile (2):
  - Providencia-Santiago
  - Temuco
- Mexico (2):
  - Zapopan, Jalisco
  - Monterrey, Nuevo León
- Puerto Rico (7):
  - Aibonito
  - Caguas
  - Ciales
  - Coto Laurel
  - Guayma
  - Guaynabo
  - Rio Piedras

REFERENCES:
- [Background] Perez A, Zhao Z, Jacks R, Spanheimer R. Efficacy and safety of pioglitazone/metformin fixed-dose combination therapy compared with pioglitazone and metformin monotherapy in treating patients with T2DM. Curr Med Res Opin. 2009 Dec;25(12):2915-23. doi: 10.1185/03007990903350011. PMID 19827910
- [Result] Perez A, Jacks R, Arora V, Spanheimer R. Effects of pioglitazone and metformin fixed-dose combination therapy on cardiovascular risk markers of inflammation and lipid profile compared with pioglitazone and metformin monotherapy in patients with type 2 diabetes. J Clin Hypertens (Greenwich). 2010 Dec;12(12):973-82. doi: 10.1111/j.1751-7176.2010.00389.x. Epub 2010 Nov 8. PMID 21122063
- See also: ACTOPLUS MET® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOPLUSMETPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 134 investigative sites in the United States (including Puerto Rico), Argentina, Chile, Guatemala, Mexico and Peru from 13 June 2007 to 29 August 2008.
Pre-assignment Details: Participants who had not received treatment with antidiabetic medication 12 weeks prior to Screening were enrolled in one of three, twice-daily (BID) treatment groups.
Groups:
- Pioglitazone 15 mg/Metformin 850 mg BID: Pioglitazone 15 mg /metformin 850 mg combination tablets, orally, twice daily for up to 24 weeks
- Pioglitazone 15 mg BID: Pioglitazone 15 mg, tablets, orally, twice daily for up to 24 weeks
- Metformin 850 mg BID: Metformin 850 mg, tablets, orally, twice daily for up to 24 weeks.
Period: Overall Study
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Started | 201 | 189 | 210
Completed | 157 | 125 | 142
Not Completed | 44 | 64 | 68

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID | Total
Number analyzed (Participants) | 201 | 189 | 210 | 600
Age Continuous [Mean (Standard Deviation); unit: years] | 54.7 (12.23) | 54.0 (12.08) | 53.7 (12.00) | 54.1 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 123 | 112 | 346
  Male | 90 | 66 | 98 | 254
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 6 | 6 | 14
  Asian | 3 | 5 | 5 | 13
  Black or African American | 12 | 13 | 14 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 123 | 109 | 124 | 356
  Multiracial | 61 | 56 | 61 | 178
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 30.84 (5.74) | 31.18 (5.50) | 30.83 (5.66) | 30.94 (5.63)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Glycosylated Hemoglobin
Description: The change between the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at final visit or week 24 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 24
Population: Participant must have baseline and at least one post-baseline value. Last Observation Carried Forward (LOCF) for missing final/week 24 visit
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 188 | 162 | 193
percentage of Glycosylated Hemoglobin | -1.83 (0.122) | -0.96 (0.131) | -0.99 (0.120)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; One-way Analysis of Covariance (ANCOVA) with treatment as a factor and the baseline value as a covariate. Least Squares (LS) mean change and LS mean of the treatment difference reported; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.86, 95% CI [0.51 to 1.22] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; One-way ANCOVA with treatment as a factor and the baseline value as a covariate. LS mean change and LS mean of the treatment difference reported; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.84, 95% CI [0.50 to 1.18] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.8919, ANCOVA; Mean Difference (Final Values) = -0.02, 95% CI [-0.37 to 0.33] — Mean Difference = Pioglitazone - metformin

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: The change between the value of Fasting Plasma Glucose collected at final visit or week 24 and Fasting Plasma Glucose collected at baseline.
Time Frame: Baseline and Week 24
Population: Participant must have baseline and at least one post-baseline value. LOCF for missing final/week 24 visit
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 196 | 176 | 202
mg/dL | -39.9 (3.48) | -22.2 (3.67) | -24.8 (3.42)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0005, ANCOVA; Mean Difference (Final Values) = 17.8, 95% CI [7.8 to 27.7] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0021, ANCOVA; Mean Difference (Final Values) = 15.1, 95% CI [5.5 to 24.7] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.5981, ANCOVA; Mean Difference (Final Values) = -2.6, 95% CI [-12.5 to 7.2] — Mean Difference = Pioglitazone - metformin

3. Secondary Outcome: Change From Baseline in Fasting Insulin
Description: The change between the Fasting Insulin value collected at final visit or week 24 and Fasting Insulin collected at baseline.
Time Frame: Baseline and Week 24
Population: Participant must have baseline and at least one post-baseline value. LOCF for missing final/week 24 visit
Measure: Least Squares Mean (Standard Error); unit: μIU/mL
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 178 | 146 | 185
μIU/mL | -3.91 (0.736) | -3.18 (0.812) | -0.98 (0.722)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.5074, ANCOVA; Mean Difference (Final Values) = 0.73, 95% CI [-1.43 to 2.88] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0047, ANCOVA; Mean Difference (Final Values) = 2.93, 95% CI [0.90 to 4.95] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0435, ANCOVA; Mean Difference (Final Values) = 2.20, 95% CI [0.06 to 4.33] — Mean Difference = Pioglitazone - metformin

4. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment - Insulin Resistance
Description: The change between Homeostasis Model Assessment of Insulin Resistance collected at final visit or week 24 and Homeostasis Model Assessment of Insulin Resistance collected at baseline. Homeostasis Model Assessment measures insulin resistance, calculated by insulin times glucose, divided by a constant (22.5).
Time Frame: Baseline and Week 24
Population: Participant must have baseline and at least one post-baseline value. LOCF for missing final/week 24 visit
Measure: Least Squares Mean (Standard Error); unit: percent of insulin resistance
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 160 | 139 | 172
percent of insulin resistance | -2.704 (0.4274) | -2.075 (0.4586) | -1.085 (0.4123)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3158, ANCOVA; Mean Difference (Final Values) = 0.629, 95% CI [-0.602 to 1.861] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0067, ANCOVA; Mean Difference (Final Values) = 1.619, 95% CI [0.452 to 2.785] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1094, ANCOVA; Mean Difference (Final Values) = 0.989, 95% CI [-0.223 to 2.201] — Mean Difference = Pioglitazone - metformin

5. Secondary Outcome: Median Percent Change From Baseline in High Sensitivity C-reactive Protein
Description: Measurement for High Sensitivity C-reactive Protein was collected at final visit or week 24 and at baseline. Percent change from baseline is calculated as: [(Week 24 - baseline levels)/baseline]*100
Time Frame: Baseline and Week 24
Measure: Median (Full Range); unit: percent
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 190 | 168 | 196
percent | -36.7 (4.6719) [-97.7 to 2060.0] | -34.0 (8.1275) [-98.9 to 2314.6] | -26.2 (12.5526) [-99.5 to 1636.3]
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; Nonparametric ANCOVA based on Tukey's normal rank transformation with a term for treatment and the baseline value as a covariate; Test type: Superiority or Other; p = 0.5963, ANCOVA; Median Difference (Final Values) = 4.88, 95% CI [-4.71 to 13.97] — The estimate of the median percent change from baseline and 95% confidence intervals were based on the Hodges-Lehmann method and the distribution-free confidence interval
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0265, ANCOVA; Median Difference (Final Values) = 12.81, 95% CI [2.88 to 22.24] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.1053, ANCOVA; Median Difference (Final Values) = 8.33, 95% CI [-1.77 to 18.07] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Change From Baseline in Adiponectin
Description: The change between Adiponectin collected at final visit or week 24 and Adiponectin collected at baseline.
Time Frame: Baseline and Week 24
Population: Participant must have baseline and at least one post-baseline value. LOCF for missing final/week 24 visit
Measure: Least Squares Mean (Standard Error); unit: mcg/ml
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 179 | 148 | 183
mcg/ml | 7.8 (0.55) | 9.2 (0.61) | -0.3 (0.55)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0806, ANCOVA; Mean Difference (Final Values) = 1.4, 95% CI [-0.2 to 3.1] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -8.1, 95% CI [-9.6 to -6.5] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -9.5, 95% CI [-11.1 to -7.9] — Mean Difference = Pioglitazone - metformin

7. Secondary Outcome: Change From Baseline in Total Cholesterol
Description: The change between Total Cholesterol collected at final visit or week 24 and Total Cholesterol collected at baseline.
Time Frame: Baseline and Week 24
Population: Participant must have baseline and at least one post-baseline value. LOCF for missing final/week 24 visit
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 178 | 154 | 182
mg/dL | 1.06 (1.183) | 4.79 (1.271) | -2.72 (1.169)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0324, ANCOVA; Mean Difference (Final Values) = 3.73, 95% CI [0.31 to 7.14] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0233, ANCOVA; Mean Difference (Final Values) = -3.78, 95% CI [-7.05 to -0.52] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -7.51, 95% CI [-10.90 to -4.12] — Mean Difference = Pioglitazone - metformin

8. Secondary Outcome: Change From Baseline in Low-Density Lipoprotein Cholesterol
Description: The change between Low-Density Lipoprotein Cholesterol collected at final visit or week 24 and Low-Density Lipoprotein Cholesterol collected at baseline.
Time Frame: Baseline and Week 24
Population: Participant must have baseline and at least one post-baseline value. LOCF for missing final/week 24 visit
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 177 | 152 | 180
mg/dL | 1.19 (2.015) | 6.08 (2.175) | -1.37 (1.998)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0993, ANCOVA; Mean Difference (Final Values) = 4.90, 95% CI [-0.93 to 10.72] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3670, ANCOVA; Mean Difference (Final Values) = -2.56, 95% CI [-8.14 to 3.01] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0119, ANCOVA; Mean Difference (Final Values) = -7.46, 95% CI [-13.26 to -1.66] — Mean Difference = Pioglitazone - metformin

9. Secondary Outcome: Change From Baseline in High-Density Lipoprotein Cholesterol
Description: The change between High-Density Lipoprotein Cholesterol collected at final visit or week 24 and High-Density Lipoprotein Cholesterol collected at baseline.
Time Frame: Baseline and Week 24
Population: Participant must have baseline and at least one post-baseline value. LOCF for missing final/week 24 visit
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 177 | 152 | 180
mg/dL | 14.20 (1.440) | 9.88 (1.552) | 6.09 (1.426)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0423, ANCOVA; Mean Difference (Final Values) = -4.31, 95% CI [-8.48 to -0.15] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -8.10, 95% CI [-12.08 to -4.12] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.728, ANCOVA; Mean Difference (Final Values) = -3.79, 95% CI [-7.93 to 0.35] — Mean Difference = Pioglitazone - metformin

10. Secondary Outcome: Change From Baseline in Triglycerides
Description: The change between Triglycerides collected at final visit or week 24 and Triglycerides collected at baseline.
Time Frame: Baseline and Week 24
Population: Participant must have baseline and at least one post-baseline value. LOCF for missing final/week 24 visit
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 180 | 157 | 184
mg/dL | -5.95 (2.901) | -5.54 (3.107) | -1.78 (2.871)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.9231, ANCOVA; Mean Difference (Final Values) = 0.41, 95% CI [-7.94 to 8.76] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3082, ANCOVA; Mean Difference (Final Values) = 4.16, 95% CI [-3.86 to 12.19] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3753, ANCOVA; Mean Difference (Final Values) = 3.75, 95% CI [-4.56 to 12.07] — Mean Difference = Pioglitazone - metformin

11. Secondary Outcome: Change From Baseline in Mean Low Density Lipoprotein Particle Concentration
Description: The change between Low Density Lipoprotein particle concentration collected at final visit or week 24 and Low Density Lipoprotein particle concentration collected at baseline.
Time Frame: Baseline and Week 24
Population: Participant must have baseline and at least one post-baseline value. LOCF for missing final/week 24 visit
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 174 | 149 | 176
nmol/L | -240.6 (23.50) | -217.2 (25.40) | -176.4 (23.36)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; One-way ANCOVA with a term for treatment and the baseline value as a covariate. LS mean change and LS mean of the treatment difference reported; Test type: Superiority or Other; p = 0.4999, ANCOVA; Mean Difference (Final Values) = 23.4, 95% CI [-44.6 to 91.4] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.0531, ANCOVA; Mean Difference (Final Values) = 64.2, 95% CI [-0.9 to 129.3] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.2369, ANCOVA; Mean Difference (Final Values) = 40.9, 95% CI [-26.9 to 108.7] — Mean Difference = Pioglitazone - metformin

12. Secondary Outcome: Change From Baseline in Mean Low Density Lipoprotein Particle Size
Description: The change between Low Density Lipoprotein collected at final visit or week 24 and Low Density Lipoprotein collected at baseline.
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Deviation); unit: nm
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 174 | 149 | 176
nm | 0.55 (0.049) | 0.6 (0.053) | 0.2 (0.049)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.5023, ANCOVA; Mean Difference (Final Values) = 0.05, 95% CI [-0.09 to 0.19] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.34, 95% CI [-0.48 to -0.21] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.39, 95% CI [-0.53 to -0.25] — Mean Difference = Pioglitazone - metformin

13. Secondary Outcome: Change From Baseline in Large Low Density Lipoprotein (L3) Concentration
Description: The change between Large Low Density Lipoprotein collected at final visit or week 24 and Large Low Density Lipoprotein collected at baseline.
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 174 | 149 | 176
nmol/L | 96.0 (12.53) | 115.7 (13.52) | 18.4 (12.46)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2849, ANCOVA; Mean Difference (Final Values) = 19.7, 95% CI [-16.5 to 55.9] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -77.6, 95% CI [-112.4 to -42.8] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -97.3, 95% CI [-133.4 to -61.2] — Mean Difference = Pioglitazone - metformin

14. Secondary Outcome: Change From Baseline in Intermediate-Density Low Density Lipoprotein Concentration
Description: The change between Intermediate-Density Low Density Lipoprotein collected at final visit or week 24 and Intermediate-Density Low Density Lipoprotein collected at baseline
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 174 | 149 | 176
nmol/L | -16.3 (3.39) | -11.0 (3.66) | -17.3 (3.37)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2894, ANCOVA; Mean Difference (Final Values) = 5.3, 95% CI [-4.5 to 15.1] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.8463, ANCOVA; Mean Difference (Final Values) = -0.9, 95% CI [-10.3 to 8.5] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2124, ANCOVA; Mean Difference (Final Values) = -6.2, 95% CI [-16.0 to 3.6] — Mean Difference = Pioglitazone - metformin

15. Secondary Outcome: Change From Baseline in Medium-Small Low Density Lipoprotein Concentration
Description: The change between Medium-Small Low Density Lipoprotein collected at final visit or week 24 and Medium-Small Low Density Lipoprotein collected at baseline
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 174 | 149 | 176
nmol/L | -63.8 (5.95) | -66.0 (6.43) | -35.3 (5.92)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.8040, ANCOVA; Mean Difference (Final Values) = -2.2, 95% CI [-19.4 to 15.0] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0008, ANCOVA; Mean Difference (Final Values) = 28.5, 95% CI [12.0 to 45.0] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0005, ANCOVA; Mean Difference (Final Values) = 30.6, 95% CI [13.4 to 47.8] — Mean Difference = Pioglitazone - metformin

16. Secondary Outcome: Change From Baseline in Small Low Density Lipoprotein Concentration
Description: The change between Small Low Density Lipoprotein collected at final visit or week 24 and Small Low Density Lipoprotein collected at baseline
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 174 | 149 | 176
nmol/L | -319.3 (28.06) | -321.3 (30.34) | -179.0 (27.91)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.9604, ANCOVA; Mean Difference (Final Values) = -2.1, 95% CI [-83.3 to 79.2] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0004, ANCOVA; Mean Difference (Final Values) = 140.3, 95% CI [62.5 to 218.0] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0006, ANCOVA; Mean Difference (Final Values) = 142.3, 95% CI [61.3 to 223.3] — Mean Difference = Pioglitazone - metformin

17. Secondary Outcome: Change From Baseline in Very Small Low Density Lipoprotein Concentration
Description: The change between Very Small Low Density Lipoprotein collected at final visit or week 24 and Very Small Low Density Lipoprotein collected at baseline
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 174 | 149 | 176
nmol/L | -255.5 (22.37) | -255.2 (24.18) | -143.8 (22.25)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.9922, ANCOVA; Mean Difference (Final Values) = 0.3, 95% CI [-64.4 to 65.1] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0004, ANCOVA; Mean Difference (Final Values) = 111.7, 95% CI [49.7 to 173.7] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0008, ANCOVA; Mean Difference (Final Values) = 111.4, 95% CI [46.8 to 175.9] — Mean Difference = Pioglitazone - metformin

18. Secondary Outcome: Change From Baseline in Mean High Density Lipoprotein Particle Concentration
Description: The change between High Density Lipoprotein collected at final visit or week 24 and High Density Lipoprotein collected at baseline.
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: μmol/L
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 174 | 149 | 176
μmol/L | 0.28 (0.271) | -0.80 (0.293) | 0.62 (0.269)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0072, ANCOVA; Mean Difference (Final Values) = -1.08, 95% CI [-1.86 to -0.29] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3682, ANCOVA; Mean Difference (Final Values) = 0.34, 95% CI [-0.41 to 1.10] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0004, ANCOVA; Mean Difference (Final Values) = 1.42, 95% CI [0.64 to 2.20] — Mean Difference = Pioglitazone - metformin

19. Secondary Outcome: Change From Baseline in Mean High Density Lipoprotein Particle Size
Description: as for outcome 18
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 174 | 149 | 176
nm | 0.15 (0.021) | 0.19 (0.022) | 0.11 (0.021)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1986, ANCOVA; Mean Difference (Final Values) = 0.04, 95% CI [-0.02 to 0.10] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1487, ANCOVA; Mean Difference (Final Values) = -0.04, 95% CI [-0.10 to 0.02] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0076, ANCOVA; Mean Difference (Final Values) = -0.08, 95% CI [-0.14 to -0.02] — Mean Difference = Pioglitazone - metformin

20. Secondary Outcome: Change From Baseline in Large High Density Lipoprotein (H4+H5) Concentration
Description: The change between Large High Density Lipoprotein collected at final visit or week 24 and Large High Density Lipoprotein collected at baseline
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: μmol/L
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 174 | 149 | 176
μmol/L | 0.70 (1.80) | 1.02 (0.194) | 0.52 (0.179)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2384, ANCOVA; Mean Difference (Final Values) = 0.31, 95% CI [-0.21 to 0.83] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.4617, ANCOVA; Mean Difference (Final Values) = -0.19, 95% CI [-0.69 to 0.31] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0593, ANCOVA; Mean Difference (Final Values) = -0.50, 95% CI [-1.02 to 0.02] — Mean Difference = Pioglitazone - metformin

21. Secondary Outcome: Change From Baseline in Intermediate-Medium High Density Lipoprotein (H3) Concentration
Description: The change between Intermediate-Medium High Density Lipoprotein collected at final visit or week 24 and Intermediate-Medium High Density Lipoprotein collected at baseline
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: μmol/L
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 174 | 149 | 176
μmol/L | 1.34 (0.285) | 1.62 (0.308) | -0.09 (0.283)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.5044, ANCOVA; Mean Difference (Final Values) = 0.28, 95% CI [-0.54 to 1.10] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0004, ANCOVA; Mean Difference (Final Values) = -1.43, 95% CI [-2.22 to -0.64] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.71, 95% CI [-2.53 to -0.89] — Mean Difference = Pioglitazone - metformin

22. Secondary Outcome: Change From Baseline in Small High Density Lipoprotein (H1+H2) Concentration
Description: The change between Small High Density Lipoprotein collected at final visit or week 24 and Small High Density Lipoprotein collected at baseline
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: μmol/L
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 174 | 149 | 176
μmol/L | -1.78 (0.349) | -3.41 (0.377) | 0.19 (0.347)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0017, ANCOVA; Mean Difference (Final Values) = -1.63, 95% CI [-2.64 to -0.62] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 1.97, 95% CI [1.01 to 2.94] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 3.60, 95% CI [2.59 to 4.61] — Mean Difference = Pioglitazone - metformin

23. Secondary Outcome: Change From Baseline in Mean Very Low Density Lipoprotein Particle Concentration
Description: The change between Very Low Density Lipoprotein collected at final visit or week 24 and Very Low Density Lipoprotein collected at baseline.
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 174 | 149 | 176
nmol/L | -2.78 (2.204) | 0.98 (2.381) | -11.30 (2.191)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2466, ANCOVA; Mean Difference (Final Values) = 3.76, 95% CI [-2.61 to 10.14] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0063, ANCOVA; Mean Difference (Final Values) = -8.52, 95% CI [-14.63 to -2.42] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -12.29, 95% CI [-18.65 to -5.93] — Mean Difference = Pioglitazone - metformin

24. Secondary Outcome: Change From Baseline in Mean Very Low Density Lipoprotein Particle Size
Description: as for outcome 23
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 174 | 149 | 176
nm | -2.64 (0.616) | -3.79 (0.666) | -0.20 (0.612)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2069, ANCOVA; Mean Difference (Final Values) = -1.15, 95% CI [-2.93 to 0.64] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0052, ANCOVA; Mean Difference (Final Values) = 2.44, 95% CI [0.73 to 4.15] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 3.59, 95% CI [1.81 to 5.36] — Mean Difference = Pioglitazone - metformin

25. Secondary Outcome: Change From Baseline in Large-Chylomicrons Very Low Density Lipoprotein Concentration
Description: The change between Large-Chylomicrons Very Low Density Lipoprotein collected at final visit or week 24 and Large-Chylomicrons Very Low Density Lipoprotein collected at baseline
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 174 | 149 | 176
nmol/L | -1.71 (0.351) | -1.97 (0.379) | -1.96 (0.349)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.6090, ANCOVA; Mean Difference (Final Values) = -0.26, 95% CI [-1.28 to 0.75] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.6169, ANCOVA; Mean Difference (Final Values) = -0.25, 95% CI [-1.22 to 0.72] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.9740, ANCOVA; Mean Difference (Final Values) = 0.02, 95% CI [-0.99 to 1.03] — Mean Difference = Pioglitazone - metformin

26. Secondary Outcome: Change From Baseline in Medium-Intermediate Very Low Density Lipoprotein (V3+V4) Concentration
Description: The change between Medium-Intermediate Very Low Density Lipoprotein collected at final visit or week 24 and Medium-Intermediate Very Low Density Lipoprotein collected at baseline
Time Frame: Baseline and Week 24
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 174 | 149 | 176
nmol/L | -4.07 (1.434) | -3.01 (1.550) | -6.48 (1.426)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.6150, ANCOVA; Mean Difference (Final Values) = 1.06, 95% CI [-3.09 to 5.21] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2346, ANCOVA; Mean Difference (Final Values) = -2.41, 95% CI [-6.38 to 1.57] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1001, ANCOVA; Mean Difference (Final Values) = -3.47, 95% CI [-7.61 to 0.67] — Mean Difference = Pioglitazone - metformin

27. Secondary Outcome: Change From Baseline in Small Very Low Density Lipoprotein (V1+V2) Concentration
Description: The change between Small Very Low Density Lipoprotein collected at final visit or week 24 and Small Very Low Density Lipoprotein collected at baseline
Time Frame: Baseline and Week 24
Population: Participant must have baseline and at least one post-baseline value. LOCF for missing final/week 24 visit
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Groups:
- Pioglitazone 15 mg/Metformin 850 mg BID: Pioglitazone 15 mg/Metformin 850 mg combination tablets, orally, twice daily for up to 24 weeks
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Number analyzed (Participants) | 174 | 149 | 176
nmol/L | 3.05 (1.249) | 5.9 (1.350) | -2.86 (1.239)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Pioglitazone 15 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1217, ANCOVA; Mean Difference (Final Values) = 2.86, 95% CI [-0.76 to 6.48] — Mean Difference = Pioglitazone & metformin - pioglitazone
Statistical Analysis 2: Comparison: Pioglitazone 15 mg/Metformin 850 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0009, ANCOVA; Mean Difference (Final Values) = -5.90, 95% CI [-9.36 to -2.44] — Mean Difference = Pioglitazone & metformin - metformin
Statistical Analysis 3: Comparison: Pioglitazone 15 mg BID vs Metformin 850 mg BID; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -8.76, 95% CI [-12.36 to -5.16] — Mean Difference = Pioglitazone - metformin

ADVERSE EVENTS:
Time Frame: Adverse events were summarized by onset date occurring on or after the first dose of double-blind study medication and on or prior to 14 days after the permanent discontinuation of the double-blind study medication.
Description: One participant was randomized to Metformin 850 mg but inadvertently received Pioglitazone 15 mg. Analyses performed on Efficacy Variables were based on Randomized Treatment; analyses on Safety Variables were based on Actual Treatment Received.
Arm/Group | Pioglitazone 15 mg/Metformin 850 mg BID | Pioglitazone 15 mg BID | Metformin 850 mg BID
Serious Adverse Events (participants affected / at risk) | 2/201 | 3/190 | 5/209
Other Adverse Events (participants affected / at risk) | 84/201 | 61/190 | 95/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone 15 mg/Metformin 850 mg BID (N=201) | Pioglitazone 15 mg BID (N=190) | Metformin 850 mg BID (N=209)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone 15 mg/Metformin 850 mg BID (N=201) | Pioglitazone 15 mg BID (N=190) | Metformin 850 mg BID (N=209)
Diarrhoea (Gastrointestinal disorders) | 18 | 5 | 32
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 7
Oedema Peripheral (General disorders) | 6 | 8 | 3
Pharyngitis (Infections and infestations) | 8 | 5 | 7
Urinary tract infection (Infections and infestations) | 6 | 5 | 9
Nasopharyngitis (Infections and infestations) | 8 | 3 | 5
Bronchitis (Infections and infestations) | 5 | 7 | 3
Glycosylated haemoglobin (Investigations) | 2 | 7 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 8 | 6
Headache (Nervous system disorders) | 11 | 5 | 10
Dizziness (Nervous system disorders) | 6 | 3 | 4
Insomnia (Psychiatric disorders) | 6 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo trial results communications up to 150 days to permit actions necessary to preserve sponsor's intellectual property. Sponsor can request changes to the results communication only for the purpose of removing non study related information that is proprietary and confidential to sponsor. Sponsor can require delay of a results communication until the study has been completed at all participating sites.